CLINICAL TRIAL: NCT00003598
Title: Retinoids and Intermediate Biomarkers for CIN II and III: Pilot Trial
Brief Title: UMCC 9609 Tretinoin in Preventing Cancer of the Cervix in Patients With Cervical Neoplasia
Acronym: IRB 1996-0189
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Dr. Mack Ruffin, University of Michigan Comprehensive Cancer Center
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000066670; P30CA046592 (NIH); CCUM-9609; NCI-P98-0131
Record Dates: First submitted 1999-11-01; First posted 2003-12-05 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Cervical Cancer; Precancerous/Nonmalignant Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tretinoin

SUMMARY:
RATIONALE: Tretinoin may help cervical neoplasia cells develop into normal cervical cells. It is not yet known whether tretinoin is more effective than a placebo in preventing cervical cancer in patients with cervical neoplasia.

PURPOSE: Randomized clinical trial to study the effectiveness of tretinoin in preventing cervical neoplasia from developing into cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether topical tretinoin reduces the number of viral genome copies of human papilloma virus (HPV) per cell and inhibits HPV E6/E7 gene expression in patients with cervical dysplasia. II. Determine the dose of tretinoin for use in a definitive trial that produces the best overall modulation of these biomarkers.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to cervical intraepithelial neoplasia classification (II vs III). Patients are randomized to 1 of 4 arms. Arm I: Patients receive low-dose tretinoin topically via cervical cap and polyurethane ether foam sponge changed daily for 4 days. Arm II: Patients receive intermediate-dose tretinoin as in arm I. Arm III: Patients receive high-dose tretinoin as in arm I. Arm IV: Patients receive placebo topically as in arm I therapy. Patients are followed for 6 months.

PROJECTED ACCRUAL: A total of 180 patients (45 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven cervical dysplasia (cervical intraepithelial neoplasia II or III) Lesions must be delineated after colposcopic biopsy No pap smears suspicious for invasive carcinoma No positive endocervical curettage

PATIENT CHARACTERISTICS: Age: Over 14 Performance status: Karnofsky 80-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Immunologic: No proliferative skin disorder (e.g., psoriasis) No diagnosed autoimmune disorders No allergy to tretinoin or latex Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception (except intrauterine device) during and for 3 months after study Normal diet with adequate protein and carbohydrate intake No in-utero exposure to diethylstilbesterol No prior malignancy No prior toxic shock syndrome

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 1 week since prior tretinoin No prior retinoids (greater than 25,000 IU vitamin A or equivalent for at least 3 months) No other tretinoin during or for 3 months after study Endocrine therapy: No concurrent regular steroids Radiotherapy: Not specified Surgery: See Disease Characteristics Other: No concurrent regular anticoagulant medication No concurrent nutritional supplements other than 2 multivitamins per day

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 1999-01; Primary Completion 2001-03 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mack T. Ruffin, MD, MPH, Study Chair — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States